CLINICAL TRIAL: NCT03671057
Title: Effectiveness Study "HospiAvontuur": Validation of a Serious Game for the Preparation of Children (4 - 6 Year Old) for a Hospital Admission for an Elective Surgical Procedure (ORL Surgery).
Brief Title: Effectiveness Study "HospiAvontuur":
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PXL University College (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PXL_hospi game
Record Dates: First submitted 2017-11-20; First posted 2018-09-14 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Children; Preoperative Anxiety; Surgery
Keywords: serious game, preoperative anxiety reduction
MeSH Terms: interventions — Midazolam; Anti-Anxiety Agents

STUDY DESIGN:
Intervention Model Description: The design of the study will be a single blinded randomized clinical trial. Children will be divided in 2 research groups: an intervention group (children who will play the game HospiAvontuur as a non-pharmacological at home preparation prior to the hospital admission. These children will not receive any pharmacological preparation - Midazolam - at the hospital) and a control group (children who do not play the game at home and do receive a pharmacological preparation - Midazolam - at the hospital). Participants will be randomly assigned to the intervention group or the control group using a computer-generated random allocation sequence, created by the study investigator (F.V.). Each patient will receive a unique randomized test number.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Two sets of cartboard boxes will be prepared. The boxes are prepared and numbered by the study investigator (F.V.) (the unique randomized test number) and distributed amongst the consultation offices of the surgeons by the researchers. To blind both the researchers and the surgeons, the 2 sets of boxes will have the same weight. The weight of the ipad is simulated in the boxes of the control group by the use of a coloring book. This will prevent patient selection bias.
  After the consultation and when the parent and the child has agreed to participate, the surgeon hands over a box to the parent. The surgeon writes the box number, name of the child, date of birth and the phone number of the child in an excel sheet. This document will be used during data procession.
  The patients participating in the trial, the treating physicians, the surgeons dispensing the study boxes, the researchers assessing outcomes and the data-managers will be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HospiAvontuur (Experimental): Intervention group - Non-pharmacological (HospiAvontuur) preparation HospiAvontuur is a simple point and click adventure game on a I-pad. The game describes the pathway which a child and his parents will take before, during and just after a hospital admission for an elective otorhinolaryngeal procedure under general anaesthesia.
  Interventions: Device: HospiAvontuur
- Midazolam (Active Comparator): control group: The children of the control group will not play the game HospiAvontuur as an at home preparation for surgery. These children will be prepared for surgery according to the current practice at the Jessa hospital. Children receive only the basic information during the consultation with the surgeon. There is no specific at home preparation required. When admitted at the hospital, children receive a pharmacological preparation, 45 - 60 minutes prior to the induction of the anaesthesia. The medication is administered orally by a small syringe in the mouth and contains Dormicum 0.3mg/kg body weight and atropine 0.02mg/kg body weight supplemented with raspberry syrup.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Device: HospiAvontuur — To be included in the study children should play the game at least one time together with one parent
  Other Names: Tablet application
  Arms: HospiAvontuur
Drug: Midazolam — current practice in Jessa
  Other Names: Anxiolytic
  Arms: Midazolam

SUMMARY:
Preoperative anxiety is frequently experienced by children undergoing anaesthesia and surgery and being separated from parents during the operation. It is associated with a significant number of adverse outcomes such as maladaptive behavioural changes and increased postoperative analgesic requirements. Pharmacological interventions such as midazolam are widely used to decrease preoperative anxiety in children. However, premedication may be associated with undesirable effects such as paradoxical reactions, prolonged sedation and adverse behavioural changes.The aim of this study is to develop and use a serious game, HospiAvontuur, which can be used during the preparation of children for an admission at the hospital. By using this game the researchers aim to reduce the usage of pharmacological interventions and to increase the use of non-pharmacological interventions, such as HospiAvontuur.

DETAILED DESCRIPTION:
The research questions for the primary outcome are formulated in 5 zero hypotheses:

Zero hypothesis 1: there is no difference in anxiety levels measured as mYPAS-SF on T1 between the two groups.

Zero hypothesis 2: there is no difference in anxiety levels measured as mYPAS-SF on T2 between the two groups.

Zero hypothesis 3: there is no difference in anxiety levels measured as ICC on T2 between the two groups.

Zero hypothesis 4: there is no difference in anxiety levels measured as VAK 4-12 on T0 between the two groups.

Zero hypothesis 5: there is no difference in change in anxiety levels measured as difference between mYPAS-SF on 2 moments (T1 versus T2) between the two groups.

The research questions for the secondary outcomes are formulated Zero hypothesis 6: there is no difference in level of emergence delirium (ED) measured during the postoperative period (T3) in the recovery room, at 4 moments, as PAED scale, between the two groups.

Zero hypothesis 7: there is no difference in level of postoperative pain measured during the postoperative period in the recovery room, as FPS-R scale and OPS scale, between the two groups.

Zero hypothesis 8: there is no difference in level of pain as FPS-R scale and problematic behaviour (PB) as modified and simplified version of the PHBQ questionnaire on day 2 and at the end of week 1 after the operation.

Design The design of the study will be a single blinded randomized clinical trial. Children will be divided in 2 research groups: an intervention group (children who will play the game HospiAvontuur as a non-pharmacological at home preparation prior to the hospital admission. These children will not receive any pharmacological preparation - Midazolam - at the hospital) and a control group (children who do not play the game at home and do receive a pharmacological preparation - Midazolam - at the hospital). Participants will be randomly assigned to the intervention group or the control group using a computer-generated random allocation sequence, created by the study investigator (F.V.). Each patient will receive a unique randomized test number.

Outcome measures As primary outcome for this research project, 2 kinds of anxiety will be measured. First the trait anxiety will be measured. Therefore the VAK 4-12 (Vragenlijst Angst Kinderen - attachment 1) will be used. To measure the state anxiety, the mYPAS-SF and the ICC will be used.

Emergence delirium: ED will be measured in the recovery room, using the five-point Pediatric Anesthesia Emergence Delirium Scale (PAED).

Pain will be measured in the recovery room, using the four-point Objective Pain Scale (OPS), at two time moments: the time of the first awaking of the child and the moment of discharge from the recovery room. For the purpose of this study, the FPS-R (Faces Pain Scale - Revised), a self-reporting pain scale, will also be used on the same time moments. This instrument will be used by a researcher.

On two time moments: 2 days after surgery and at the end of the first week after surgery, parents will receive a phone call from one of the doctors from the anesthesia department or the study investigator.

Both postoperative pain and problematic behaviour will be questioned during a semi-structured interview. The FPS-R will be used for pain measurement and 10 questions will be asked in order to get a good impression of the child's postoperative behaviour (table 1).

One version of the FPS-R will be handed over to the parents and the child at the moment of discharge from the hospital. Parents will be informed that they can expect a phone call from a researcher or an anesthesia staff member and that some questions including the pain perception will be asked.

Power analysis

Based on the duration of the research project, the expected subjects that could be included in the study, the controlling of the variables and based on previous research from Marechal et al (2016), the following power analysis was calculated:

A total research population of 164 subjects (82 subjects per group), would be required to demonstrate a 8 point difference in m-YPAS score at time of induction (level of significance of p < 0.05 and power of 80%). The mean mYPAS score at time of induction, after MDZ premedication in the study of Marechal et al (2016) was 43.74 (SD = 18.32).

Data received from the OR database (1/12/2015 - 30/11/2016) show that approximately 300 children undergo ORL surgery over 12 months. Our study will start at 01/09/2017 and will end on 31/05/2018 (a period of 9 months). During this period approximately 225 children will be operated in the OR. As surgeons are able to set parents at ease to participate in the study because no harm will done to the child and since children nor parents won't notice the presence of the researcher in the OR (performing the observations), it is expected that most parents and children will participate. However, some parents are not keen on scientific studies. Others will not be interested in participating because their mind is set on the child that needs surgery rather than on other things. Moreover, the number of children undergoing ORL surgery is not always constant and there is also a risk of loss-to-follow-up. Therefore, the sample size of 164 patients will be inflated to 90 participants per group (180 in total) to account for a possible 10% loss-to-follow-up.

Statistics The significance of the differences between the two groups for the scores of VAK4-12, mYPas at T1, mTPAS at T2, ICC will be tested with Mann-Whitney U-tests. The significance of the differences between T2 and T1 for the two groups will be measured with two-way ANOVA. All statistical analyses will be done in the package SAS.

Ethics During the recruiting of the participants it is important that both parents and children are fully informed about the randomization process. In general, playing a serious game is considered to be a pleasant activity and children who are assigned to the intervention group may consider themselves to be lucky. On the other hand parents may think that playing a game and therefore not receiving the standard pharmacological treatment may be considered as unfavourable. When providing information to parents it is crucial to make it clear that both the non-pharmacological as the pharmacological strategies have a scientific basis and that no harm will be done to the children.

The non-pharmacological preparation of children before surgery is considered standard procedure in many hospitals. At the Jessa Hospital this is not yet the case although questions about this issue have been risen some time ago, according to the anaesthesia department. At this moment there is no specific non-pharmacological alternative in use. Therefore this research project could be an answer to this issue. The results from the study could support the decision in whether a non-pharmacological preparation program could be introduced.

During the observations of the children in the preoperative holding area and in the operating room during anesthesia induction, it is possible that the researcher or the anesthesiologist can happen to hear some information from the child or the parent about gaming experiences. This can be the case when the child recognizes specific information in the OR that he/she has experienced during the gameplay. When this is the case, the researcher and/or the anesthesiologist should make a remark on the observation form. Even if this is the case, the objective observation and scoring on the scale should continue as planned.

ELIGIBILITY:
Inclusion Criteria:

* Children from 4 up to (and included) 7 years old. The children represent a large group within the otorhinolaryngeal discipline and these children are within the same cognitive phase when it comes to playing a serious game
* Children who need otorhinolaryngeal surgery for the first time.
* Children and at least one of the parents are able to comprehend and speak the Dutch language.
* Children who will receive a mask induction of the anaesthesia.

Exclusion Criteria:

* Older and younger children than the mentioned age group.
* Children who do not have a complete comprehension of the Dutch language. Children will not be excluded based on cultural or background information.
* Children who had previous surgical experiences both elective or urgent.
* The following children will also be excluded from participation: children with mental retardation, children that have had opioids or sedative during the past month, children with early birth, children with behavioural dysfunction and children with a delayed cognitive development.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 164 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
mYPAS-SF (pre-operative) | At baseline: at the beginning of the preoperative process
  For the measurement of the state anxiety, the mYPAS-SF (attachment 3) (modified Yale Preoperative Anxiety Scale - Short Version) will be used. In previous research projects usually the mYPAS (attachment 4) is used. The mYPAS was developed in 1995 (Kain et al, 1995) and modified in 1997 (Kain et al, 1997). It has been used in more than 100 studies spanning diverse health fields, such as anesthesia, surgery, paediatrics and dentistry (Cuzzocrea et al, 2013; Davidson et al, 2006; Huet et al, 2011; Weldon et al, 2004; Fortier et al, 2009; Fortier et al, 2010). This measurement instrument uses 5 items, each representing a different domain of child anxiety, and is used at 4 points in time during the preoperative phase. These 4 time points are: preoperative holding, walk to the OR, entrance to the OR (child enters the OR but has not yet seen the anesthesia mask), and introduction to the anesthesia mask (Jenkins et al, 2014).

SECONDARY OUTCOMES:
VAK 4-12 (Vragenlijst Angst Kinderen) for anxiety (pre-operative) | Up to two weeks before baseline measurement: the VAK4-12 will be completed at home, before any intervention has taken place.
  In order to determine any baseline imbalances between the research groups, the VAK4-12 questionnaire will be used. The VAK4-12 (Vragenlijst Angst Kinderen) is a Dutch questionnaire to determine the level of subjective experienced fear in children of 4-6 years old (trait anxiety). It is a reconstructed version of the Revised Fear Survey Schedule for Children. The scale offers scores on 5 subscales and can be completed by children and their parent(s) together. It is a scale which is easy to complete and takes about 20 minutes. In scientific research this questionnaire can be used to select anxious and non-anxious children. It can also be used in effectiveness studies for interventions which focus on anxiety reduction.
ICC (pre-operative) | At baseline: at the beginning of the preoperative process
  The ICC (Induction Compliance Checklist) is an observational checklist for describing the compliance of a child towards the induction of general anaesthesia. The checklist consists of 11 items which indicate the compliance. The ICC score is the sum of the items checked. A perfect induction, during which the child does not show negative behaviors, fear or anxiety is scored as 0. This instrument was developed by the research group of Kain et al (1998).
PAEDS (Pediatric Anxiety Emergency delirium Scale) (post-operative) | Immediately after surgery
  The PAED (Pediatric Anesthesia Emergence Delirium Scale) is an observational checklist for describing emergence delirium in the postoperative phase. The scale incorporates cognitive and agitation assessment items and is generally acknowledged to be the most valid and reliable. A score of 10 or above has the highest diagnostic sensitivity and specificity (Bong CL, Ng AS, 2009; Janseen NJ, Tan EY, Staal M, et al, 2011).
OPS (Objective Pain Score) (Post-operative) | Immediately after surgery
  The OPS (Objective Pain Score) is an observational scale for postoperative pain measurement. The scale is a good stand-alone tool to scale pain and to ascertain the need for analgesia and is a good tool to refer to when the NRS is indicative of mild or moderate pain (Tandom M. et al, 2016). At this moment the scale is the standard used instrument in the recovery room.
Faces Pain Scale - Revised (FPS-R) (post-operative) | After 2 days and after 1 week of surgery
  The Faces Pain Scale - Revised (FPS-R) (Hicks CL, von Baeyer CL, Spafford P., et al, 2001) is a self-report measure of pain intensity developed for children. It was adapted from the Faces Pain Scale (Bieri D., Reeve R., Champion GD., et al., 1990) to make it possible to score the sensation of pain on the widely accepted 0-to-10 metric. The scale shows a close linear relationship with visual analog pain scales across the age range of 4-16 years. It is easy to administer and requires no equipment except for the photocopied faces.

CONTACTS AND LOCATIONS:
Overall Officials: Annemie IF Spooren, PhD, Principal Investigator — PXL University College
Locations (1):
- Jessa, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided